CLINICAL TRIAL: NCT06780410
Title: A Phase III Clinical Study to Evaluate the Efficacy, Tolerability, and Safety of Bempedoic Acid in Patients with Hyperlipidemia Not Adequately Controlled by Statins
Brief Title: A Clinical Study to Evaluate the Efficacy, Tolerability, and Safety of Bempedoic Acid
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gan & Lee Pharmaceuticals. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BDP-HLD-301
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Primary Hyperlipidemia
Keywords: Bempedoic Acid; Hyperlipidemia; Efficacy; Safety
MeSH Terms: conditions — Hyperlipidemias | interventions — 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bempedoic acid (Experimental): Once daily
  Interventions: Drug: Bempedoic Acid Tablet
- Placebo (Placebo Comparator): Once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bempedoic Acid Tablet — Once daily, oral
  Arms: Bempedoic acid
Drug: Placebo — Once daily, oral
  Arms: Placebo

SUMMARY:
This trial is a phase III study to evaluate the efficacy , tolerability, and safety of Bempedoic Acid Tablets in patients with hyperlipidemia not adequately controlled by Statins.

ELIGIBILITY:
Inclusion Criteria:

* 1. 18 years and older, male or female.
* 2. 18 kg/m2 ≤Body Mass Index (BMI) ≤35 kg/m2.
* 3. Participants must agree to use reliable contraception from the screening day until 30 days after the last dose, and must not donate sperm or eggs for assisted reproduction purposes.
* 4. Fully understand the purpose and requirements of the study, voluntarily participate in the clinical trial, and sign a written informed consent form, capable of completing the entire study process.

Exclusion Criteria:

* 1. Known allergy to any component of the investigational drug or its excipients, or a history of allergic diseases (e.g., asthma, urticaria, eczema) or allergic constitution.
* 2. Fasting triglycerides (TG) ≥ 5.64 mmol/L (≥ 500 mg/dL) at screening.
* 3. History of malignant tumors prior to screening.
* 4. History of drug, alcohol, amphetamines, or other drug abuse.
* 5. Participation in other clinical studies and use of other investigational drugs or medical devices within 3 months prior to screening or within 5 half-lives of the drugs (whichever is longer).
* 6. Pregnant or breastfeeding females, or those with a positive human chorionic gonadotropin (HCG) pregnancy test.
* 7. Any other factors that the investigator believes makes the participant unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Percentage change from baseline in LDL-C levels at Week 12 | Baseline, Week 12

SECONDARY OUTCOMES:
Percentage change from baseline in total cholesterol (TC) levels at Week 12 | Baseline, Week 12
Adverse events (AEs) and serious adverse events (SAEs) during the study | Baseline, Week 13

CONTACTS AND LOCATIONS:
Locations (1):
- Site 01, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided